CLINICAL TRIAL: NCT06795087
Title: Discharge Medication Use Post-Operatively in GU Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00121391; LCI-GU-PO-NMC-001 (Other: Atrium Health)
Record Dates: First submitted 2025-01-24; First posted 2025-01-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Genitourinary Cancer
Keywords: Genitourinary Cancer; Cystectomies; Nephrectomies; Prostatectomies
MeSH Terms: conditions — Urogenital Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Education Cohort
- Post-Education Cohort
  Interventions: Other: Opioid Medication Disposal Education

INTERVENTIONS:
Other: Opioid Medication Disposal Education — Education on opioid medication disposal will be provided in the form of a pamphlet created by Atrium Health based on FDA resources and will be given to all participants at discharge (cystectomy, nephrectomy, prostatectomy) beginning in the second year, approximately 13 months from when the first participant is enrolled or until a minimum of 100 evaluable participants are enrolled in the pre-education cohort, whichever occurs last.
  Groups: Post-Education Cohort

SUMMARY:
The main purpose of this research study is to determine the amount of opioids that are taken after discharge following a cystectomy, nephrectomy (partial or total), or prostatectomy surgeries via a 30-day post- discharge opioid use and disposal survey. We will also evaluate the impact of an opioid disposal education pamphlet on proper disposal of unused opioids.

DETAILED DESCRIPTION:
This prospective, non-therapeutic trial aims to evaluate the amount of prescribed opioid medications GU cancer patients are consuming post-discharge following surgical procedure of cystectomies, nephrectomies, and prostatectomies.

Enrolled participants will complete a 30-day post-discharge survey evaluating the usage of prescribed opioids and opioid disposal habits, as well as a patient satisfaction survey. Furthermore, participants will be offered to complete an optional CAHPS® Surgical Care Survey to assess patients' experiences with surgical care during in hospital stay and outpatient office visits.

Education on opioid medication disposal will be provided in the form of a pamphlet to participants that are enrolled beginning in year 2 (approximately month 13) from when the first participant is enrolled or after a minimum of 100 evaluable participants are enrolled in the pre-education cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information.
2. Age ≥ 18 years at the time of enrollment
3. Scheduled to undergo surgical cystectomy, partial or total nephrectomy or prostatectomy for a cancer diagnosis.
4. Ability to read and understand the English and/or Spanish language.
5. As determined by the enrolling investigator, ability of the participant to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants ≥ 18 years of age or older who will undergo planned cystectomy, nephrectomy (partial or total), or prostatectomy for a GU cancer diagnosis will be approached to enroll into the study.
Sampling Method: Non-Probability Sample
Enrollment: 684 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Discharge opioids consumed in 30 days after discharge | 30 days after discharge
  For each participant who was prescribed an opioid medication after urology surgery, the number of opioid pills consumed in 30 days after discharge will be captured as a categorical variable from the "Opioid Use and Disposal Survey". Participant-reported options include None, About one-fourth of all pills, About half of all pills, About three-fourths of all pills, or All. Participants who report that they received an opioid prescription but did not fill it will be captured as taking None.

SECONDARY OUTCOMES:
Number of participants filling opioid prescription | 30 days after discharge
  For each participant who was prescribed an opioid medication after urology surgery, whether or not the prescription was filled will be reported as a binary variable on the "Opioid Use and Disposal Survey".
Participant-reported reasons for not filling opioid prescription | 30 days after discharge
  For each participant who reported not filling their opioid prescription, reason for not filling the prescription will be captured on the "Opioid Use and Disposal Survey". Options include: Pain was controlled without taking any opioid medications, Concern about side effects, Concern about developing addiction or dependence, Other (explain).
Participant-reported reasons for not taking all pills | 30 days after discharge
  For each participant who reported filling their opioid prescription but did not take all of their pills, reason for not taking all of the prescribed pills will be captured on the "Opioid Use and Disposal Survey". Options include: Pain was controlled without taking all pills, Side effects were too severe, Concern about developing addiction or dependence, Other (explain).
Participant-reported pain control after discharge | 30 days after discharge
  Each participant will report what their average daily pain score was in the first week after discharge on the "Opioid Use and Disposal Survey". This will be reported on a scale of 0 - 10, with 0 indicating "no pain" and 10 indicating "worst possible pain".
Number of participants receiving a refill after discharge | 30 days after discharge
  For each participant who was prescribed an opioid medication after urology surgery, whether or not the participant received a refill of opioid medication(s) during the 30-day period post-discharge will be captured as a binary variable from the electronic medical records.
Participant-reported disposal method for left-over opioids | 30 days after discharge
  For each participant who filled the opioid prescription that they received, the method of disposal or storage of excess opioid medication will be captured as a categorical variable on the "Opioid Use and Disposal Survey". The possible methods include: Threw away in trash, Stored in an unlocked cabinet, Stored in a locked cabinet, Flushed down the toilet, Brought to a pharmacy or hospital, Brought to a law enforcement center, Still taking prescribed opioids, Other (explain)
Patient Satisfaction Survey Item 1 - "I would recommend this institution to a friend or family for treatment." | 30 days after discharge
  The satisfaction level with surgery will be captured for each participant from a single administration of a study-specific "Patient Satisfaction Survey" that contains 5 items and is administered 30 days after discharge. This item will be measured for each participant with 5-point Likert scale response options (Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree).
Patient Satisfaction Survey Item 2 - "The staff provided adequate information and education prior to discharge regarding my recovery at home (ex. wound care and pain management)." | 30 days after discharge
  The satisfaction level with surgery will be captured for each participant from a single administration of a study-specific "Patient Satisfaction Survey" administered 30 days after discharge. This item will be measured for each participant with 5-point Likert scale response options (Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree).
Patient Satisfaction Survey Item 3 - "Prior to my discharge, I or my caregiver clearly understood the timing and purpose for taking each of my medications." | 30 days after discharge
  The satisfaction level with surgery will be captured for each participant from a single administration of a study-specific "Patient Satisfaction Survey" administered 30 days after discharge. This item will be measured for each participant with 5-point Likert scale response options (Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree).
Patient Satisfaction Survey Item 4 - "During the hospital stay, nurses and doctors treated me with courtesy and respect." | 30 days after discharge
  The satisfaction level with surgery will be captured for each participant from a single administration of a study-specific "Patient Satisfaction Survey" administered 30 days after discharge. This item will be measured for each participant with 5-point Likert scale response options (Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree).
Patient Satisfaction Survey Item 5 - "Following prostatectomy, I preferred to be discharged the same day." | 30 days after discharge
  The satisfaction level with surgery will be captured for each participant from a single administration of a study-specific "Patient Satisfaction Survey" administered 30 days after discharge. This item will be measured for each participant with a 7-level categorical response (Strongly Agree, Agree, Neither Agree nor Disagree, Disagree, Strongly Disagree, I did not have prostatectomy, I had a prostatectomy however, I was not discharged the same day).
CAHPS Surgical Care Survey - Number of patients with top-box ratings of preparation for surgery | 30 days after discharge
  From the CAHPS Surgical Care Survey, a binary variable will indicate whether or not the participants reported a top-box response for questions in the "preparation for surgery" domain. Response options include: Yes, definitely (top-box); Yes somewhat; No
CAHPS Surgical Care Survey - Number of patients with top-box ratings of preoperative communication | 30 days after discharge
  From the CAHPS Surgical Care Survey, a binary variable will indicate whether or not the participants reported a top-box response for questions in the "preoperative communication" domain. Response options include: Yes, definitely (top-box); Yes somewhat; No
CAHPS Surgical Care Survey - Number of patients with top-box ratings of day of surgery attentiveness | 30 days after discharge
  From the CAHPS Surgical Care Survey, a binary variable will indicate whether or not the participants reported a top-box response for questions in the "day of surgery attentiveness" domain. Response options include: Yes (top-box); No
CAHPS Surgical Care Survey - Patients' rating of surgeon | 30 days after discharge
  From the CAHPS Surgical Care Survey, patient-reported rating of their surgeon on a scale of 0 to 10, with 0 being the worst and 10 being the best.
CAHPS Surgical Care Survey - Patients' rating of anesthesiologist | 30 days after discharge
  From the CAHPS Surgical Care Survey, patient reported rating of their anesthesiologist on a scale of 0 to 10, with 0 being the worst and 10 being the best.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Riggs, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States